CLINICAL TRIAL: NCT06709157
Title: Immunocompetent Versus Immunocompromised Tuberculosis (TB) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer of Medical Microbiology and Immunology, Sohag University
Other Study IDs: Soh-Med-24-08--05PD
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis
Keywords: HIV; immunocompromised; cytokines
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: P24 antigens and antibody — estimation of antigens and antibodies to diagnose HIV
Diagnostic Test: zeihl - Nelsen stain — staining sputum from patients with HIV to detect tubercle bacilli
Diagnostic Test: culture on Lowenstein jensen media — spenciem will be inoculated on LJ media and kept for 2-8 weeks, to see small white colonies
Diagnostic Test: Molecular detection of antibiotic resistance — to see the pattern of antibiotic resistance of tubercle bacilli

SUMMARY:
Tuberculosis (TB) is caused by Mycobacterium tuberculosis and is one of the top 10 causes of mortality worldwide. It is estimated that in 2017, 10 million people were infected with TB, and 1.6 million died from the disease, including 0.3 million people with human immunodeficiency virus (HIV) infection . TB remains the primary killer of HIV-positive individuals. TB incidence is falling at about 2% per year . Airborne transmission of M. tuberculosis typically causes TB infection in both immunocompetent and immunocompromised hosts and the disease is symptomatic and contagious .

DETAILED DESCRIPTION:
TB and HIV infections are strictly linked together. TB is the most common opportunistic infection and causes high morbidity rate among people living with HIV. Because of the decrease in cell-mediated immunity, HIV alters the pathogenesis of TB, thereby expressively increasing the risk of TB in HIV-positive patients and eventually leading to more severe complications and forms of TB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic chest disease

Exclusion Criteria:

* Patients with other respiratory or infectious diseases.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: This prospective study will be conducted on 100-200 patients with pulmonary and extra pulmonary TB attending Sohag University Hospital during the period from September 2024 to August 2025
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The Prevalance of tubercuolsis in immunocompetent patients suffereing from chronic chest problems | December 2024- June 2025
  Patients suffering from chronic chest problems will be screened for presence of TB bacilli using chest X-ray, sputum smear, culture on LJ media, detection of DNA of TB bacilli using PCR
The prevalence of tuberculosis in HIV patients | December 2024- June 2025
  Detection of tubercle bacilli in HIV positive patients , these patients will be screened for presence of TB bacilli using chest X-ray, sputum smear, culture on LJ media, detection of DNA of TB bacilli using PCR

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Shafik, Lecturer, Principal Investigator — Sohag university, Faculty of medicine; Asmaa T Mostafa, Lecturer, Study Chair — Sohag university, Faculty of Medicine; Ebtisam M Gad, Lecturer, Study Chair — Sohag university, Faculty of Medicine; Mona M Abdelrahman, Lecturer, Study Chair — Sohag university, Faculty of Medicine; Dina H Mohamed, Lecturer, Study Chair — Sohag university, Faculty of medicine
Locations (1):
- Faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No